CLINICAL TRIAL: NCT01804855
Title: An Investigation of the Clinical Effectiveness of Adolescent Weight-management Delivered Via a Portable Device
Brief Title: Effectiveness of a Smartphone App for Adolescent Obesity Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's University Hospital, Ireland (Other)
Collaborators: University College Cork (Other); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TSCUH-2013-1158
Record Dates: First submitted 2013-03-04; First posted 2013-03-05 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Obesity; Impaired Health; Psychosocial Problem; Physical Activity; General Nutrition Disorder
Keywords: Obesity; mobile health; telemedicine; family-based treatment
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- W82GO (Active Comparator): Usual face-to-face care as per the W82GO multidisciplinary treatment intervention (phase 1 for 6 weeks and phase 2 for 46 weeks).
  Interventions: Behavioral: W82GO
- Smartphone (Experimental): Usual care for Phase 1 of treatment. Treatment during Phase 2 of intervention using the Reactivate smartphone application only.
  Interventions: Device: smartphone application

INTERVENTIONS:
Behavioral: W82GO — MDT delivered obesity intervention integrating behavioural change methods in order to reduce obesity; improve nutrition; increase physical activity; improve sleep; reduce sedentarism and increase self-esteem
  Arms: W82GO
Device: smartphone application — Behavior change smartphone application for adolescents aiming to reduce obesity
  Other Names: Reactivate application
  Arms: Smartphone

SUMMARY:
Though face-to-face treatment of childhood obesity can be effective, it is time consuming and costly. This study will test whether treatment can be delivered via an Android app and whether such treatment reduces obesity.

ELIGIBILITY:
Inclusion Criteria:

* child aged between 12.0 and 17.0 years,
* child BMI =/> 98th percentile,
* first language is English (or fluent in English)
* parent/s willing to participate in the programme with their child
* completion of written informed consent and/or assent prior to any study-specific procedures

Exclusion Criteria:

* severe intellectual difficulties,
* obesity secondary to genetic condition,
* limitations to engaging in physical activity
* use of medication known to effect body weight;
* limitations to using a smartphone device
* known family issues that would affect general compliance and attendance at follow-up visits.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 126 (Estimated)
Dates: Start 2013-02 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
BMI Z score | 12 months
  Z score calculated using LMS growth software

SECONDARY OUTCOMES:
Body Fat Mass | 12 months
  Measured using Tanita Bioelectric impedance analyser
Physical activity | 12 months
  Measured using Geneactive acclerometery
Laboratory tests | 12 months
  Lipids; glucose; insulin; HbA1C; liver function
Psychosocial health | 12 months
  Measured using the Child Behaviour Check list
Safety | 12 months
  Adverse effects will be monitored throughout the study and a full report at 12 months will be given.

CONTACTS AND LOCATIONS:
Overall Officials: Grace O'Malley, MSc BSc, Principal Investigator — Temple Street Children's University Hospital; Amanda Burls, MD, PhD, Study Chair — University of Oxford; Sinead Murphy, MD, Study Chair — Temple Street Children's University Hospital; Ivan Perry, MD, PhD, Study Director — University College Cork
Locations (1):
- Temple Street Children's University Hospital, Dublin, Ireland

REFERENCES:
- [Background] O'Malley G, Brinkley A, Moroney K, McInerney M, Murphy S, Kileen S, Murphy N. Establishing a hospital based obesity service: An Irish Experience. Obesity Facts 2012;5(S10):9.
- [Background] O'Malley G, Brinkley A, Moroney K, McInerney M, Murphy S, Kileen S, Murphy N. Is the Temple Street W82Go Healthy Lifestyles Programme effective in reducing BMI SDS?. Obesity Facts 2012;5(S10):223
- [Derived] Tully L, Sorensen J, O'Malley G. Pediatric Weight Management Through mHealth Compared to Face-to-Face Care: Cost Analysis of a Randomized Control Trial. JMIR Mhealth Uhealth. 2021 Sep 14;9(9):e31621. doi: 10.2196/31621. PMID 34519665
- [Derived] O'Malley G, Clarke M, Burls A, Murphy S, Murphy N, Perry IJ. A smartphone intervention for adolescent obesity: study protocol for a randomised controlled non-inferiority trial. Trials. 2014 Jan 31;15:43. doi: 10.1186/1745-6215-15-43. PMID 24485327
- See also: Website for W82GO programme and trial — http://w82go.ie
- See also: Website for Temple Street Children's University Hospital — http://cuh.ie